CLINICAL TRIAL: NCT06136234
Title: COVE (Caring for Vets and Service Members)
Brief Title: Caring for Vets and Service Members: Caring Contacts for Stressed and Distressed Veterans and Service Members
Acronym: COVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Face the Fight (Unknown)
Responsible Party: Principal Investigator, Kate Comtois, Professor: School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00019011
Record Dates: First submitted 2023-10-23; First posted 2023-11-18 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Stress; Distress, Emotional
Keywords: suicidal ideation; suicide cognitions
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: All outcome measures are completed by the participant via online survey.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental Condition with intensive assessment (Experimental): Caring Contacts plus best available resources, with monthly EMAs during study year
  Interventions: Behavioral: Caring Contacts; Behavioral: Best Available Resources Alone
- Control Condition with intensive assessment (Active Comparator): Best available resources, with monthly EMAs during study year
  Interventions: Behavioral: Best Available Resources Alone
- Experimental Condition without intensive assessment (Experimental): Caring Contacts plus best available resources, without monthly EMAs during study year
  Interventions: Behavioral: Caring Contacts; Behavioral: Best Available Resources Alone

INTERVENTIONS:
Behavioral: Caring Contacts — Caring Contacts are brief, periodic messages sent over 1 year that express unconditional care and concern
  Arms: Experimental Condition with intensive assessment; Experimental Condition without intensive assessment
Behavioral: Best Available Resources Alone — Participants will be offered information about best available resources and will receive an email summarizing the resources with links and contact information. These resources are tailored to best serve the participant based on information they share during the online survey or during conversations with study staff.

SUMMARY:
The goal of this clinical trial is to study stressed or distressed veterans and service members. Researchers will compare Caring Contacts plus best available resources to best available resources alone to see if reduces distress and prevents thoughts of suicide.

DETAILED DESCRIPTION:
The objective of this study is to evaluate whether Caring Contacts via text message are beneficial to veterans and service members experiencing stress or distress. In the past, Caring Contacts interventions have focused on individuals who are already suicidal and not a more general population. In addition, a core objective of this study is to understand the mechanisms of action of Caring Contacts and thus has included an ecological momentary assessment (EMA) component that will allow us to determine when and how Caring Contacts is making an impact.

Study aims are to

Evaluate if stressed or distressed veterans receiving Caring Contacts are at greater or less risk of suicidal ideation or behavior as evidenced by:

Decreased mean and reduction in variability of indicators of suicide risk (motivation to live, passive ideation, active ideation, suicide intent, and urges to harm self) acquired during Ecological Momentary Assessment periods.

Reduced risk of suicidal ideation (HASS-I) and cognitions (SCS-R) during follow-up.

Examine diverse veterans' experiences with Caring Contacts (i.e., access, satisfaction, preferences, potential mechanisms)

Evaluate if veterans receiving Caring Contacts will show a decrease in distress (i.e., isolation, depression, substance use, loneliness, defeat, hopelessness, and psychological pain)

Identify potential mechanisms of action for Caring Contacts by exploring the relationship between potential mechanisms (i.e., mattering, connectedness, social responsibility, and entrapment), distress, and suicide risk observed during ecological momentary assessment periods to identify potential mechanisms of action of Caring Contacts on decreasing distress and suicide risk

ELIGIBILITY:
Inclusion Criteria:

* US service member or veteran
* 18 years or older
* Lives in the United States
* Stressed (recent separation from or in transition out of the military, unemployment, financial strain, unhoused, or suicide loss, etc.) or distressed (isolation, depression, substance use, loneliness, defeat, hopelessness, psychological pain, or suicidal ideation, etc.)
* Willingness to be contacted periodically by text message and either email or postal mail

Exclusion Criteria:

- Unable to consent due to inability to understand the consent form due to cognitive limitations or insufficient English (as determined by inability to pass the consent quiz items)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Suicide risk Visual Analog Scales (VAS) | 3 EMA assessments/day for 14 days at baseline; then either 3 EMA assessments/day for 7 days at 12 months OR 3 EMA assessments/day for 7 days/month for 12 months (depending on EMA condition)
  Suicide risk indicators rated on Visual Analog Scales (VAS; 0-10) acquired during Ecological Momentary Assessment periods. Core constructs of suicide risk selected and worded to maximize face validity: motivation to live, passive ideation, active ideation, and urges for suicide. Higher scores indicate higher suicidal risk (motivation to live is reverse coded).
Suicidal Ideation | Baseline and 12 month follow-up
  Harkavy-Asnis Suicide Scale (HASS-I), adapted version for study procedures. Min=0, max=60, higher scores indicate higher suicidal ideation.
Suicide Cognitions | Baseline and 12 month follow-up
  Suicide Cognitions Scale - Revised, Min=16, max=80, higher scores indicate more suicidal cognitions.

SECONDARY OUTCOMES:
Experience of receiving Caring Contacts | 12 month follow-up
  Participants will be asked to describe their experiences with Caring Contacts via an online survey and a qualitative interview with a subset of participants
Depression | Baseline and 12 month-up
  Patient Health Questionnaire-9 (PHQ-9), Min=0, max=30, higher scores indicate higher degree of depression severity.
Substance Abuse | Baseline and 12 month follow-up
  Short Inventory of Problems - Alcohol and Drugs (SIP-AD)
Loneliness | Baseline and 12 month follow-up
  NIH Loneliness Scale, Min=5, max=25, higher scores indicate increased loneliness.
Defeat | Baseline and 12 month follow-up
  The Defeat Scale, Min=0, max=64, higher scores indicate greater defeat.
Hopelessness | Baseline and 12 month follow-up
  Beck's Hopelessness Scale (BHS), Min=0, max=20, higher scores indicate greater hopelessness.
Psychological Pain | Baseline and 12 month follow-up
  Unbearable Psychache Scale-3 (UPS-3), Min=3, max=15, higher scores indicate greater psychological pain.

OTHER OUTCOMES:
Potential Mechanism: Entrapment | 3 EMA assessments/day for 14 days at baseline; then either 3 EMA assessments/day for 7 days at 12 months OR 3 EMA assessments/day for 7 days/month for 12 months (depending on EMA condition)
  A single item, "I feel trapped," acquired during Ecological Momentary Assessment periods. Min=1, max=7, higher score indicates increased feelings of entrapment.
Potential Mechanism: Personal and Social Responsibility | 3 EMA assessments/day for 14 days at baseline; then either 3 EMA assessments/day for 7 days at 12 months OR 3 EMA assessments/day for 7 days/month for 12 months (depending on EMA condition)
  Responsibility Scale acquired during Ecological Momentary Assessment periods. Min=8, max=40, higher scores indicate greater sense personal and social responsibility.
Potential Mechanism: Mattering | 3 EMA assessments/day for 14 days at baseline; then either 3 EMA assessments/day for 7 days at 12 months OR 3 EMA assessments/day for 7 days/month for 12 months (depending on EMA condition)
  General Mattering Scale acquired during Ecological Momentary Assessment periods. Min=5, max=20, higher scores indicate greater sense of mattering.
Potential Mechanism: Perceived Burdensomeness | 3 EMA assessments/day for 14 days at baseline; then either 3 EMA assessments/day for 7 days at 12 months OR 3 EMA assessments/day for 7 days/month for 12 months (depending on EMA condition)
  A single item, "I felt that I was a burden to other people, or that they would be better off without me," acquired during Ecological Momentary Assessment periods. Min=1, max=7, higher score indicates increased feelings of burdensomeness.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Comtois, PhD/MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will only make de-identified data and associated documentation available to users outside the research team under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Wright B, Evanson A, Casey C, Law KC, Rogers AH, Comtois KA. Exploring the Impact of the Caring Contacts Intervention on the Stress and Distress of Veterans and Service Members: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Aug 13;14:e72140. doi: 10.2196/72140. PMID 40801426